CLINICAL TRIAL: NCT04171102
Title: Neo-neurogenesis in 3D Dynamic Responsive Implant for Inguinal Hernia Repair PorFlor
Brief Title: Neo-nervegenesis in Inguinal Hernia Implant ProFlor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Giuseppe Amato, Consultant Professor, University of Cagliari
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Neo-nervegenesis in ProFlor
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Inguinal Hernia
Keywords: Hernia implants; Biologic response; Neo-nervegenesis; Regenerative scaffold
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Short term post inguinal hernia repair wit ProFlor (Active Comparator): Determining presence and level of maturation of nervous structures in the hernia implant named ProFlor at 3-5 weeks post implantation
  Interventions: Device: ProFlor Hernia implant
- Mid term post inguinal hernia repair wit ProFlor (Active Comparator): Determining presence and level of maturation of nervous structures in the hernia implant named ProFlor at 3-4 months post implantation
  Interventions: Device: ProFlor Hernia implant
- Long term post inguinal hernia repair wit ProFlor (Active Comparator): Determining presence and level of maturation of nervous structures in the hernia implant named ProFlor at 6-8 months post implantation
  Interventions: Device: ProFlor Hernia implant

INTERVENTIONS:
Device: ProFlor Hernia implant — Inguinal hernia repair

SUMMARY:
The investigation is aimed at specifically demonstrating the ingrowth of newly formed nervous elements within a 3D dynamic responsive implant for inguinal hernia repair.

DETAILED DESCRIPTION:
Biopsy specimen were excised at defined postoperative stages from patients who underwent hernia repair with the 3D prosthesis named ProFlor. Scope of the study was to determine the presence, quantity and quality of the neural ingrowth within the implant fabric. Histology revealed the presence of multiple nerve clusters that, starting from the early stage post-implantation, increased in number and degree of maturation. In the long term, neural elements assumed the typical aspect of normal nervous structures complete in all components. The development of highly specialized tissue such as nerves, together with other components of the abdominal wall already described in literature, seems to finalize a regenerative response. This kind of behavior, being the expected result from a device intended for the cure of inguinal hernia and its degenerative source, seems to be coherent with the pathogenesis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent inguinal hernia repair with the prosthetic device named ProFlor
* Patients undergoing recurrent inguinal hernia repair after primary repair with the prosthetic device named ProFlor
* Patients undergoing surgical procedure in the groin area after inguinal hernia repair with the prosthetic device named ProFlor

Exclusion Criteria:

* Patients who underwent inguinal hernia repair with conventional flat meshes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Amato, MD, Principal Investigator — University of Cagliari

IPD SHARING:
Plan to Share IPD: Yes
Tissue specimen and histological records upon request
Time Frame: from actual date until december 2021
Access Criteria: personal contact

REFERENCES:
- [Background] Amato G, Lo Monte AI, Cassata G, Damiano G, Romano G, Bussani R. A new prosthetic implant for inguinal hernia repair: its features in a porcine experimental model. Artif Organs. 2011 Aug;35(8):E181-90. doi: 10.1111/j.1525-1594.2011.01272.x. Epub 2011 Jul 13. PMID 21752035
- [Background] Amato G, Romano G, Agrusa A, Marasa S, Cocorullo G, Gulotta G, Goetze T, Puleio R. Biologic response of inguinal hernia prosthetics: a comparative study of conventional static meshes versus 3D dynamic implants. Artif Organs. 2015 Jan;39(1):E10-23. doi: 10.1111/aor.12416. PMID 25626584
- [Background] Amato G, Romano G, Puleio R, Agrusa A, Goetze T, Gulotta E, Gordini L, Erdas E, Calo P. Neomyogenesis in 3D Dynamic Responsive Prosthesis for Inguinal Hernia Repair. Artif Organs. 2018 Dec;42(12):1216-1223. doi: 10.1111/aor.13286. Epub 2018 Oct 14. PMID 30318605
- [Result] Amato G, Agrusa A, Puleio R, Calo P, Goetze T, Romano G. Neo-nervegenesis in 3D dynamic responsive implant for inguinal hernia repair. Qualitative study. Int J Surg. 2020 Apr;76:114-119. doi: 10.1016/j.ijsu.2020.02.046. Epub 2020 Mar 10. PMID 32169570

RESULTS

PARTICIPANT FLOW:
Groups:
- Neonervegenesis in ProFlor Hernia Implant in the Short Term: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 3-5 weeks post-implantation
- Neonervegenesis in ProFlor Hernia Implant in the Mid Term: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 3-4 months post-implantation
- Neonervegenesis in ProFlor Hernia Implant in the Long Term: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 6-8 months post-implantation
Period: Overall Study
Arm/Group | Neonervegenesis in ProFlor Hernia Implant in the Short Term | Neonervegenesis in ProFlor Hernia Implant in the Mid Term | Neonervegenesis in ProFlor Hernia Implant in the Long Term
Started | 4 | 5 | 6
Completed | 4 | 5 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Inguinal hernia patients operated with ProFlor who needed further surgery in the previously operated groin for various pathologies
Groups:
- Short Term Post-implantation: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 3-5 weeks post-implantation
- Mid Term Post-implantation: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 3-4 months post-implantation
- Long Term Post-implantation: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 6-8 months post-implantation
- Total: Total of all reporting groups
Arm/Group | Short Term Post-implantation | Mid Term Post-implantation | Long Term Post-implantation | Total
Number analyzed (Participants) | 4 | 5 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 11
  >=65 years | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (4561) | 59.6 (4871) | 61.5 (4881) | 58.23 (4581)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 5 | 6 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 4 | 5 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Ingrowth of Newly Formed Nervous Elements Within Hernia Implant ProFlor
Description: Post-operative assessment of neonervegenesis within hernia implant ProFlor at short, mid and long term post-implantation
Time Frame: 3 weeks until 8 months post-implantation
Population: Patients who underwent inguinal hernia repair with ProFlor
Measure: Mean (Standard Deviation); unit: μm^2
Groups:
- Short Term Post Implantation: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 3-5 weeks post implantation
- Mid Term Post Implantation: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 3-4 months post implantation
- Long Term Post-implantation: Determining presence and level of maturation of nervous structures in the hernia implant ProFlor at 6-8 months post implantation
Arm/Group | Short Term Post Implantation | Mid Term Post Implantation | Long Term Post-implantation
Number analyzed (Participants) | 4 | 5 | 6
μm^2 | 999.75 (113.32) | 1044 (695.95) | 2094 (490.82)
Statistical Analysis 1: Comparison: Short Term Post Implantation vs Mid Term Post Implantation vs Long Term Post-implantation; Test type: Other; p = 0.028, t-test, 2 sided — <0.05

ADVERSE EVENTS:
Time Frame: 1 year
Description: All participant underwent biopsy from the implanted prosthesis. Being the prosthesis positioned in the inguinal area outside of the abdominal cavity, this minimally invasive procedure produces no risks of mortality. Also risks for serious adverse events are nullified because the tissue removal do not involve any vital organs
Arm/Group | Short Term Post-implantation | Mid Term Post-implantation | Long Term Post-implantation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No